CLINICAL TRIAL: NCT00289042
Title: The Use of Enoxaparin Compared to Unfractionated Heparin for Short Term Antithrombotic Therapy in Atrial Fibrillation Patients Undergoing TEE Guided Cardioversion: Assessment of Cardioversion Using Transesophageal Echocardiography (ACUTE) II Randomized Multicenter Study
Brief Title: Assessment of Cardioversion Using Transesophageal Echocardiography II (ACUTE II)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2879
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2005-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial thrombus; cardioversion; enoxaparin; low molecular weight heparin; transesophageal echocardiography
MeSH Terms: conditions — Atrial Fibrillation | interventions — Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
SPECIFIC AIM: To test the safety and feasibility of using low molecular weight heparin (LMWH, enoxaparin sodium; Lovenox, Sanofi-Aventis) in lieu of unfractionated heparin (UFH) as antithrombotic therapy for patients in atrial fibrillation undergoing transesophageal echocardiography (TEE) guided chemical or electrical cardioversion to sinus rhythm.

HYPOTHESIS: Early cardioversion from atrial fibrillation can be safely performed using a short-term anticoagulation strategy of low molecular weight heparin (Lovenox, Sanofi-Aventis) compared to unfractionated heparin, accompanied by a TEE examination prior to cardioversion. The use of LMWH with TEE will result in a safe, cost-effective, and possible efficacious approach to cardioversion of atrial fibrillation compared to UFH with TEE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic or paroxysmal atrial fibrillation of > 2 days duration who are candidates for early chemical or electrical cardioversion
* Patients with atrial flutter with a documented history (electrocardiography) of atrial fibrillation
* Males and females 18 years of age or older
* Patients have available results of routine clinical labs for standard clinical chemistry and complete blood count within the previous 14 days

Exclusion Criteria:

* An INR > 1.4 in patients who have received warfarin prior to enrollment.
* Use of IV heparin for more than 72 hours immediately prior to randomization.
* Patients with contraindications to TEE, such as dysphagia, or esophageal strictures.
* Patients who will need anticoagulation discontinued because of elective intervening procedure, such as cardiac catheterization or surgery.
* Patients with contraindications to warfarin or heparin
* Patients who require concomitant therapy during the study period with any drug known to affect coagulation or platelet function (i.e. ASA, NSAID, antiplatelet drugs)
* Women of childbearing potential, unless pregnancy can be excluded by medical history incompatible with pregnancy or by serum or urine beta HCG levels.
* Patients who are hemodynamically unstable and thus may require immediate cardioversion.
* Weight less than 40 kg (88 pounds) or more than 125 kg (275 pounds)
* History of gastrointestinal bleeding disorder and/or endoscopically verified ulcer disease within the last year
* History of intracranial or retinal bleeding, or other known disorders with an increased risk of bleeding
* Ischemic stroke in the previous three months
* Uncontrolled hypertension (systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Malignancy currently under active treatment, including melanoma
* Patients with renal insufficiency (creatinine > 2.0 mg/dL) or are renal transplant subjects
* Patients with anemia (Hgb less than 10 gm/dL)
* Patients with thrombocytopenia (platelet count less than 100 x 10^9/L)
* Positive fecal hemoglobin test
* Life expectancy of less than 6 months
* History of drug and/or alcohol abuse within the last two years
* Patients unable or unwilling to give informed consent
* Patients unable or unwilling to return for follow-up
* Prisoners or wards of the state
* Patients with psychological problems that may decrease compliance with the protocol
* Not willing to complete the Quality of Life Questionnaires x 3
* Participating in another clinical trial and/or taking an investigational medication in the past 30 days
* Patient language, learning skills, or home environment unconducive to self-management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1999-12; Study Completion 2004-11

PRIMARY OUTCOMES:
ischemic stroke
transient ischemic attack
peripheral embolism
major or minor bleeding
death
length of stay (LOS)
return to normal sinus rhythm (NSR)

SECONDARY OUTCOMES:
quality of life
cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Allan L. Klein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Klein AL, Grimm RA, Murray RD, Apperson-Hansen C, Asinger RW, Black IW, Davidoff R, Erbel R, Halperin JL, Orsinelli DA, Porter TR, Stoddard MF; Assessment of Cardioversion Using Transesophageal Echocardiography Investigators. Use of transesophageal echocardiography to guide cardioversion in patients with atrial fibrillation. N Engl J Med. 2001 May 10;344(19):1411-20. doi: 10.1056/NEJM200105103441901. PMID 11346805
- [Background] Murray RD, Deitcher SR, Shah A, Jasper SE, Bashir M, Grimm RA, Klein AL. Potential clinical efficacy and cost benefit of a transesophageal echocardiography-guided low-molecular-weight heparin (enoxaparin) approach to antithrombotic therapy in patients undergoing immediate cardioversion from atrial fibrillation. J Am Soc Echocardiogr. 2001 Mar;14(3):200-8. doi: 10.1067/mje.2001.109505. PMID 11241016
- [Background] Murray RD, Shah A, Jasper SE, Goodman A, Deitcher SR, Katz WE, Malouf JF, Stoddard MF, Grimm RA, Klein AL; ACUTE II pilot study. Transesophageal echocardiography guided enoxaparin antithrombotic strategy for cardioversion of atrial fibrillation: the ACUTE II pilot study. Am Heart J. 2000 Jun;139(6):E1-7. doi: 10.1067/mhj.2000.106628. PMID 10827367
- [Derived] Elliott DJ, Zhao L, Jasper SE, Lieber EA, Klein AL, Weintraub WS. Health status outcomes after cardioversion for atrial fibrillation: results from the Assessment of Cardioversion Using Transesophageal Echocardiography (ACUTE) II Trial. Am Heart J. 2008 Aug;156(2):374.e1-6. doi: 10.1016/j.ahj.2008.05.008. PMID 18657673